CLINICAL TRIAL: NCT01675141
Title: Lenalidomide Maintenance Therapy in Multiple Myeloma: A Phase II Clinical and Biomarker Study
Brief Title: Lenalidomide Maintenance Therapy for Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Original investigator left the NIH and the primary outcome was not reached
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Dickran Kazandjian, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120192; 12-C-0192
Record Dates: First submitted 2012-08-25; First posted 2012-08-29 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Multiple Myeloma
Keywords: NK Cell Function; Immunomodulatory Drugs; T Cell Activity; Immune Stimulatory Effects; Extended Dosing
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lenalidomide Maintenance Therapy for Multiple Myeloma (Experimental): 10 mg oral daily, on days 1-21 of repeated 28 day cycles, to continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — 10 mg oral daily, on days 1-21 of repeated 28 day cycles, to continue until disease progression or unacceptable toxicity.

SUMMARY:
Background:

* Multiple myeloma is rarely curable, but it is treatable. Initial treatment is directed at controlling symptoms and reducing the number of myeloma cells. It continues until the cancer stops responding to treatment. At that time, treatment may switch to maintenance therapy, which is given to try to extend the response of the first therapy for as long as possible. Research suggests that lenalidomide maintenance therapy may delay the time for myeloma cells to start to grow and possibly improve survival.
* Lenalidomide is a drug that may reduce or prevent the growth of cancer cells. Researchers want to look at the long-term effect of lenalidomide on immune cells. It will also look at the effects of extended treatment on the cancer and the immune system.

Objectives:

- To test the long-term effectiveness of lenalidomide therapy for multiple myeloma.

Eligibility:

- Individuals at least 18 years of age with newly diagnosed or relapsed multiple myeloma.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine sample will be collected. A bone scan and bone marrow biopsy will also be performed.
* Participants will receive lenalidomide maintenance treatment. It will be given according to the standard of care for multiple myeloma. Participants will take lenalidomide every day for 21 days of repeated 28-day cycles.
* Treatment will be monitored with frequent blood tests. Blood tests will look at the effect of the treatment on the immune system.
* Treatment will continue as long as the cancer does not worsen and the side effects are not severe.

DETAILED DESCRIPTION:
Background:

Multiple myeloma (MM) remains largely an incurable disease with an estimated median survival of 6-7 years in standard risk myeloma and 2-3 years in high risk disease despite treatment with autologous stem cell transplantation (ASCT).

Maintenance therapy to achieve sustained suppression of residual disease following chemotherapy or ASCT has long been viewed as a desirable approach for extending survival in MM.

Giving the immunomodulatory drug lenalidomide after induction or re-induction treatment may stimulate the immune system in various ways to stop or slow the return of cancer.

It is not yet known how immune stimulatory effects of extended dosing with lenalidomide in the maintenance setting correlate with clinical benefits.

Objectives:

Assess T cell (cluster of differentiation 4 (CD4), cluster of differentiation 8 (CD8), natural killer T cell (NKT) and normal killer (NK) cell numbers in peripheral blood during the

course of lenalidomide maintenance therapy in treated MM patients.

Eligibility:

Patients with multiple myeloma who have achieved stable disease or better response, assessed at greater than or equal to 4 weeks after completing induction or re-induction treatment

Age greater than or equal to 18 years

Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-2

Adequate hematological parameters defined by: absolute neutrophil count greater than or equal to 1.0 K/microL, hemoglobin greater than or equal to 8 g/dL, and platelet count greater than or equal to 75 K/microL

Adequate hepatic function, with bilirubin < 1.5 times the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times ULN

Adequate renal function with creatinine clearance (CrCl) of greater than or equal to 40 mL/min. CrCl will be calculated using the Cockcroft-Gault method. If the calculated CrCl based on Cockcroft-Gault method is <40 mL/min, patient will have a 24 hr urine collection to measure CrCl. The measured CrCl must also be greater than or equal to 40 ml/min

Design:

Single arm, single stage, phase II trial of lenalidomide maintenance for treated MM patients who have stable or responsive disease.

After screening, eligibility determination, and enrollment; subjects will receive lenalidomide 10 mg by mouth daily on days 1-21 of repeated 28-day cycles. When necessary, lenalidomide will be held and restarted in accordance with accepted clinical dose modification guidelines.

Subjects may continue lenalidomide until disease progression or unacceptable toxicity or completion of two years of lenalidomide therapy and the 30 day safety follow-up visit.

Blood will be obtained to assess changes in T cell (CD4, CD8), NKT and NK cell numbers by flow-cytometric analysis at pre-specified time points during lenalidomide maintenance.

Blood samples and/or bone marrow samples where possible, will be used for additional research studies, which may include functional analyses of immune-cell subsets, analyses for cytokines, chemokines, antibodies, tumor cell antigen targets, and/or other markers.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with multiple myeloma treated with induction therapy or re-induction therapy, who at the time of study enrollment have documented evidence of stable disease response or better according to International Myeloma Workshop Consensus Panel. The response assessment must occur at least 4 weeks after completion of their last treatment.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of lenalidomide in patients
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Patient must have adequate hematologic, renal, hepatic, and cardiac function as defined by:

  * Absolute neutrophil count greater than or equal to 1.0 K/microL independent of growth factor support
  * Platelets greater than or equal to 75K/microL
  * Hemoglobin greater than or equal to 8 g/dL (transfusions are permissible)
  * Calculated creatinine (CrCl) clearance of greater than or equal to 40 mL/min. using the Cockcroft-Gault method. If the calculated CrCl based on Cockcroft-Gault method is
  * Total bilirubin less than or equal to 1.5 mg/dL, aspartate aminotransferase (AST)/ serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/ serum glutamic-pyruvic transaminase (SGPT) less than or equal to 3 times ULN
* Females of childbearing potential (FCBP) must agree to use two effective forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study. The two methods of effective contraception must include one highly effective method (i.e. intrauterine device (IUD), hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom, diaphragm, cervical cap). FCBP must be referred to a qualified provider of contraceptive methods if needed.
* A FCBP is defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* A FCBP must have two negative serum or urine pregnancy tests prior to starting study drug. The first pregnancy test must be performed within 10-14 days prior to the start of study drug and the second pregnancy test must be performed within 24 hours prior to prescribing the study drug. The prescriptions of study drug must be filled within 7 days.
* Male patients must agree to use a latex condom during sexual contact with FCBP while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a successful vasectomy.
* Patient must be able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation. Patients intolerant to acetylsalicylic acid (ASA) may use warfarin or low molecular weight heparin.
* Patient must understand and voluntarily sign an informed consent form, with the understanding that the patient may withdraw consent at any time without prejudice to future medical care.

EXCLUSION CRITERIA:

* Patients with progressive or refractory multiple myeloma (MM), as defined by International Myeloma Workshop Consensus Panel criteria.
* Refractory to lenalidomide in the most recent line of therapy, as defined by the International Myeloma Consensus Panel criteria - as failure to achieve minimal response or development of progressive disease while on lenalidomide or within 30 days of lenalidomide therapy
* Patients who are receiving any other investigational agents with the intent to treat myeloma. Permitted concurrent therapies include:
* Bisphosphonates
* Radiotherapy to single stable disease site
* Plasma cell leukemia
* Pregnant or lactating females. Because there is a potential risk for adverse events to nursing infants secondary to treatment of the mother with lenalidomide, lactating females must agree not to breast feed while taking lenalidomide.
* Uncontrolled hypertension or diabetes
* Active hepatitis B or C infection
* Diagnosed or treated for another malignancy within 3 years prior to study enrollment, with the exception of complete resection of non-melanoma skin cancer, or an in situ malignancy
* Previous diagnosis of another malignancy with any evidence of residual disease.
* Patients seropositive for the human immunodeficiency virus (HIV), and/or those who are taking anti-retroviral treatment for HIV/acquired immune deficiency syndrome (AIDS)
* Prior organ transplant requiring immunosuppressive therapy
* Prior allogeneic stem cell transplant
* Patients requiring continuous, systemic immunosuppressive therapy
* Patients with myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled cardiac arrhythmias, or electrocardiographic evidence of acute ischemia
* Patients with conditions that would prevent absorption of the study drug
* Uncontrolled intercurrent illness including but not limited to uncontrolled infection or psychiatric illness/social situations that would compromise compliance with study requirements
* Significant neuropathy greater than or equal to Grade 3 at baseline
* Contraindication to concomitant anticoagulation prophylaxis
* Major surgery within 1 month prior to enrollment
* Patients who were previously exposed and who developed severe adverse events, hypersensitivity or desquamating rash to either thalidomide or lenalidomide

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-08-20 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2017-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dickran Kazandijicn, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kyle RA, Rajkumar SV. Multiple myeloma. N Engl J Med. 2004 Oct 28;351(18):1860-73. doi: 10.1056/NEJMra041875. No abstract available. PMID 15509819
- [Background] Landgren O, Kyle RA, Pfeiffer RM, Katzmann JA, Caporaso NE, Hayes RB, Dispenzieri A, Kumar S, Clark RJ, Baris D, Hoover R, Rajkumar SV. Monoclonal gammopathy of undetermined significance (MGUS) consistently precedes multiple myeloma: a prospective study. Blood. 2009 May 28;113(22):5412-7. doi: 10.1182/blood-2008-12-194241. Epub 2009 Jan 29. PMID 19179464
- [Background] Rajkumar SV, Kyle RA. Multiple myeloma: diagnosis and treatment. Mayo Clin Proc. 2005 Oct;80(10):1371-82. doi: 10.4065/80.10.1371. PMID 16212152
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0192.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide Maintenance Therapy for Multiple Myeloma
Started | 11
Completed | 0
Not Completed | 11
Not completed — Lenalidomide outside NIH | 3
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 4
Not completed — No treatment, per protocol | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide Maintenance Therapy for Multiple Myeloma
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.05 (8.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 1
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic | 9
  Mexican, Cuban, Puerto Rican, Central/So. American | 2
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Longitudinal Assessment of T Cell (Cluster of Differentiation 4 (CD4), Cluster of Differentiation 8 (CD8), Natural Killer T-cell (NKT) and Natural Killer (NK) Cell Counts
Description: Peripheral blood samples will be collected to assess T cell (CD4, CD8), NKT and NK cell counts using flow cytometry.
Time Frame: participants were followed for the duration of their treatment, an average of 2 years
Population: This outcome was not done because this study was closed prior to full enrollment. Given study closure, the primary endpoint could not be and was not evaluated. There was not an adequate amount of specimens collected to arrive to any analyses conclusions.
Arm/Group | Lenalidomide Maintenance Therapy for Multiple Myeloma
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the number of serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 37 months and 12 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide Maintenance Therapy for Multiple Myeloma
Number analyzed (Participants) | 11
Participants | 11

3. Secondary Outcome: Duration of Response
Description: Duration of response is defined as time from response to disease progression or death. Progression is assessed by the International Myeloma Workshop Consensus Panel Criteria. Progressive disease requires any one or more of the following: increase of ≥25% from baseline or lowest response value in Serum M component, Urine M component, free light chain or bone marrow plasma cell percentage. Lowest response value does not need to be a confirmed value. Serum M-component absolute increase must be ≥0.5 g/dl. The serum M-component increases of ≥1 gm/dl are sufficient to define relapse if starting M-component is ≥5 g/dl. Urine M-component absolute increase must be ≥200mg/24h. Only in patients without measureable serum and urine M-protein levels: the absolute increase in difference between involved and uninvolved free light chain levels must be >10mg/dl.
Time Frame: participants were followed for the duration of their treatment, an average of 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide Maintenance Therapy for Multiple Myeloma
Number analyzed (Participants) | 10
Months | NA [0.9 to NA] — The median and upper limit of 95% CI is NR (not reached). The median and upper limit were not reached because there was not enough follow up time to reach a median or upper limit.

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from study entry until progression or death. Progression is assessed by the International Myeloma Workshop Consensus Panel Criteria. Progressive disease requires any one or more of the following: increase of ≥25% from baseline or lowest response value in Serum M component, Urine M component, free light chain or bone marrow plasma cell percentage. Lowest response value does not need to be a confirmed value. Serum M-component absolute increase must be ≥0.5 g/dl. The serum M-component increases of ≥1 gm/dl are sufficient to define relapse if starting M-component is ≥5 g/dl. Urine M-component absolute increase must be ≥200mg/24h. Only in patients without measureable serum and urine M-protein levels: the absolute increase in difference between involved and uninvolved free light chain levels must be >10mg/dl.
Time Frame: participants were followed for the duration of their treatment, an average of 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide Maintenance Therapy for Multiple Myeloma
Number analyzed (Participants) | 11
months | NA [16.2 to NA] — The median and upper limit of 95% CI is NR (not reached). The median and upper limit were not reached because there was not enough follow up time to reach a median or upper limit.

5. Secondary Outcome: Natural Killer (NK) Cell Function and Activity
Description: Percent of target cell lysis by NK cells
Time Frame: participants were followed for the duration of their treatment, an average of 2 years
Population: as for outcome 1
Arm/Group | Lenalidomide Maintenance Therapy for Multiple Myeloma
Number analyzed (Participants) | 0

6. Secondary Outcome: Changes in B Cell Subsets, Myeloid Derived Suppressor Cells and T Regulatory Cells by Phenotypic Analysis During the Course of Therapy
Description: Percent change in total number of B Cell Subsets, Myeloid Derived Suppressor Cells and T Regulatory Cells by Phenotypic Analysis During the Course of Therapy
Time Frame: participants were followed for the duration of their treatment, an average of 2 years
Population: as for outcome 1
Arm/Group | Lenalidomide Maintenance Therapy for Multiple Myeloma
Number analyzed (Participants) | 0

7. Secondary Outcome: Expression of Cereblon (CRBN) and How it Relates to Natural Killer (NK) Cell Number and Activity
Description: Relative fold change in CRBN and correlation (R2) to NK cell number and activity.
Time Frame: participants were followed for the duration of their treatment, an average of 2 years
Population: as for outcome 1
Arm/Group | Lenalidomide Maintenance Therapy for Multiple Myeloma
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 37 months and 12 days
Arm/Group | Lenalidomide Maintenance Therapy for Multiple Myeloma
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide Maintenance Therapy for Multiple Myeloma (N=11)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (6)
Alkaline phosphatase increased (Investigations) | 4 (6)
Anemia (Blood and lymphatic system disorders) | 5 (11)
Aspartate aminotransferase increased (Investigations) | 4 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (3)
CPK increased (Investigations) | 3 (6)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Creatinine increased (Investigations) | 5 (11)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 1 (1)
Edema face (General disorders) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 2 (3)
Fever (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 2 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (6)
Infections and infestations - Other, dental abscess (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 8 (18)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, primary prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neutrophil count decreased (Investigations) | 8 (25)
Pain (General disorders) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Platelet count decreased (Investigations) | 4 (9)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
White blood cell decreased (Investigations) | 10 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT01675141/Prot_SAP_000.pdf
  • Informed Consent Form (2014-06-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT01675141/ICF_001.pdf